

**Project Title**: Patient Priorities Care (PPC) for older Adults with Multiple Chronic Conditions Achieved through Primary and Specialty Care Alignment; **Principal Investigator**: Ardeshir Hashmi, MD (phone: 216-445-4415)

# **Patient Study Information Sheet**

Thank you for taking the time to review this information.

This information sheet gives you information about the study, which the study staff will then review with you. The study staff will explain the purpose of the study, any risks to you and what is expected of you. You are free to ask questions about the study at any time. This study was developed by a research team at Yale University, and has been approved by Cleveland Clinic's Institutional Review Board. Before you learn more about the study, it is important for you to know that your participation in this study is entirely voluntary. You may decide not to take part in, or to withdraw from, the study at any time.

## Why are you being asked to participate in this study?

You are being asked to participate in this study because you are an older adult with multiple health conditions who receives care at a Cleveland Clinic primary care department at one of our Family Health Centers in Lakewood or Brunswick.

### What is the purpose of this study?

The primary objective of this study is to help researchers learn about a new approach to patient care called: *Patient Priorities Care*. We are asking health care providers to try discussing the information collected in different ways, to see what works best for older adults with more than one health problem.

Researchers plan to interview/survey patients like you to ask some health-related questions in an effort to help learn about this new approach.

### What are the requirements and time commitment to participate?

You are being asked to participate in two 15-minute interviews/surveys (one to be conducted in the near future and one to be conducted in about 9 months from now). The interviews/surveys may be conducted over the phone or in person.

If you agree, the interview/survey will involve questions about your health, the type of help you get from your healthcare team, and how you feel about your health care as well as what is burdensome (difficult).

There are no right or wrong answers to any of these questions. Everyone feels differently about their health and their health care. That is why we are asking a lot of people, including you, so we can get a general idea of the range of people's thoughts.

# What are the benefits to taking part in this study?

You will experience no direct benefit from participating in this study. Although this study will not benefit you personally, we hope that our results will add to the knowledge about how doctors/health care providers can provide the best possible care to their patients.

### Are there any risks to you in participating in this study?

There are no known or anticipated risks to you for participating.

The study team will gather information from the Cleveland Clinic electronic medical record about the people who participate in this interview/survey including their health, number of medications, and number of healthcare/doctor visits. This information will be combined and reported as a group



**Project Title**: Patient Priorities Care (PPC) for older Adults with Multiple Chronic Conditions Achieved through Primary and Specialty Care Alignment; **Principal Investigator**: Ardeshir Hashmi, MD (phone: 216-445-4415)

and it will be entirely de-identified after the identifying code is destroyed. De-identified data will be shared with the Yale University research team.

All of your interview/survey responses will be held in confidence and will not be shared with your doctor/health care providers. Only the researchers involved in this evaluation and those responsible for research oversight will have access to the information you provide as part of this interview/survey. Your responses will be numbered and the code linking your number with your name will be stored in a separate database. After all the interviews/surveys are complete, the code will be destroyed so your interview/survey is de-identified.

As with all studies, there is a potential risk of loss of confidentiality of your data. Every effort will be made to keep your information confidential through the use of the following safeguards: All data will be stored in a password-protected and encrypted (hidden) database accessible only by the research team. Participant names will be replaced by study number so that all others receiving data will not be able to connect a name with data. Only unique study identification numbers will identify participants in research databases. All data will be reported in aggregate (combined as a group) and will not be linked to specific individuals.

### Do I have to participate in the research?

Your participation is strictly voluntary. Your decision to participate will not impact your current or future medical care a Cleveland Clinic, nor will it affect your relationship with your doctor or health care providers.

You may choose not to take part or may leave the study at any time. Leaving the study will not result in any penalty or loss of compensation.

#### What other options are there?

Your participation is strictly voluntary. The alternative is to not participate.

#### What are the costs?

There are no costs for you to participate.

You will receive in the mail/or in person a \$10.00 gift card for participating in each of the study interviews.

The IRS requires CCF to report payments to an individual of \$600 or greater (in a calendar year) on a Form 1099-MISC. Your name, address and social security number will be collected to track the payments made to you and, if you receive \$600 or greater, will be used to process a Form 1099-MISC.

#### Who do I contact if I have questions about the research?

If you have questions about the study before or after you have agreed, you may ask the study coordinators Toyomi Goto (216-444-8424) or Jackie Fox, RN (216-444-4590) for assistance at any time or you can contact Dr. Ardeshir Hashmi (principal investigator) at 216-445-4415. If you have any questions about your rights as a research subject, you can contact the Institutional Review Board at (216) 444-2924.

Participation in the interview/survey will indicate your agreement to participate in the research.